CLINICAL TRIAL: NCT07157384
Title: Randomized Controlled Trial Comparing REMIssion of Type 2 Diabetes Between Intermittently Scanned Continuous Glucose Monitoring and Capillary Blood Glucose Monitoring When Added to Low-calorie Meal Replacement and Diabetes Self-management Education: The REMIT2D isCGM Trial
Brief Title: REMIssion of Type 2 Diabetes Between Intermittently Scanned Continuous Glucose Monitoring and Capillary Blood Glucose Monitoring When Added to Low-calorie Meal Replacement and Diabetes Self-management Education
Acronym: REMIT2D isCGM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Collaborators: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REMIT2D isCGM
Record Dates: First submitted 2025-08-07; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
Keywords: low-calorie meal replacement; remission; intermittently scanned continuous glucose monitoring; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- isCGM + LCMR + DSME (Experimental): Group using an intermittently scanned continuous glucose monitor and receiving low calorie meal replacement and diabetes self management education
  Interventions: Dietary Supplement: Low calorie meal replacement plan; Behavioral: Diabetes self management education; Device: Intermittently scanned continuous glucose monitoring
- CBG + LCMR + DSME (Active Comparator): Group using a capillary blood glucose monitor and receiving low calorie meal replacement and diabetes self management education
  Interventions: Dietary Supplement: Low calorie meal replacement plan; Behavioral: Diabetes self management education; Device: capillary blood glucose monitoring

INTERVENTIONS:
Dietary Supplement: Low calorie meal replacement plan — intervention provided to both arms in 2 out of the 3 study phases: Phase 1 (total dietary replacement) and Phase 2 (food re-introduction)
Behavioral: Diabetes self management education — intervention provided to both arms throughout study conducted as in-person session and telephone sessions
Device: Intermittently scanned continuous glucose monitoring — intervention provided to the intervention arm only: isCGM + LCMR + DSME
  Arms: isCGM + LCMR + DSME
Device: capillary blood glucose monitoring — intervention provided to the control arm only: CBG + LCMR + DSME
  Arms: CBG + LCMR + DSME

SUMMARY:
The goal of the study is to evaluate the effectiveness of intermittently scanned continuous glucose monitoring compared to capillary blood glucose monitoring among people with type 2 diabetes initiating low calorie meal replacement plus diabetes self-management education in improving the proportion of patients achieving remission of type 2 diabetes. This is an open-label randomized controlled trial with 2 treatment arms randomized in a 1:1 manner.

The Investigators hypothesize that the use of intermittently scanned continuous glucose monitoring will improve the percentage of participants achieving remission of type 2 diabetes (remission to prediabetes or remission to normoglycemia), among adults with type 2 diabetes starting low calorie meal replacement and diabetes self-management education compared to a control group using capillary blood glucose monitoring at 18-30 weeks follow-up (end of Phase 2).

The primary outcome of the study is to compare the percentage of participants who achieve remission of type 2 diabetes (remission to prediabetes with HbA1c 6.0% to 6.4% or remission to normoglycemia with HbA1c < 6.0% using no antihyperglycemic agents for ≥ 3 consecutive months) at 18-30 weeks follow-up between intermittently scanned continuous glucose monitoring vs. capillary blood glucose monitoring, when combined with low calorie meal replacement and diabetes self-management education.

Participants in both arms complete 3 phases of the study. Phase 1: total dietary replacement, Phase 2: food re-introduction and Phase 3: remission, while receiving diabetes self-management education sessions over a span of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old
* T2D treated with ≤ 3 non-insulin antihyperglycemic agents
* A clinical diagnosis of T2D for > 6 months and ≤ 6 years ago
* HbA1c 6.0-9.0% on 2 or 3 antihyperglycemic agents, HbA1c 6.5-9.0% on 1 antihyperglycemic agent, or HbA1c 7.0-9.0% on 0 antihyperglycemic agents
* BMI 27-44.9 kg/m2
* Not currently using a real-time CGM or isCGM
* Willing to adhere to LCMR and initiate isCGM or CBG monitoring, and capable to do so as judged by investigator

Exclusion Criteria:

* Current or prior use of insulin (except for prior management of gestational diabetes mellitus)
* Are pregnant or breastfeeding, or planning to become pregnant in the next 2 years
* Severe or progressive retinopathy
* Have a history of cardiovascular disease: coronary artery disease (CAD): prior myocardial infarction, previous unstable angina, documented CAD on angiography with stenosis >50%, imaging evidence of myocardial ischemia, coronary revascularization), peripheral arterial disease (lower extremity stenosis exceeding 50%, previous limb angioplasty, stenting or bypass surgery; or previous limb or foot amputation due to circulatory insufficiency or ankle brachial index of < 0.9 in at least one limb.), cerebrovascular disease (history of ischemic or hemorrhagic stroke or > 50% carotid stenosis), or heart failure
* Chronic kidney disease with estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m2 or eGFR 60-90 ml/min/1.73 m2 with urine albumin to creatinine ratio (uACR) > 20 mg/mmol (any previously resolved macroalbuminuria will be considered as a reason for ineligibility, at the investigator's discretion)
* Active binge eating disorder or other eating disorder
* Uncontrolled mental health disorder
* Current use of atypical antipsychotic or corticosteroid
* Use of other implanted medical devices, such as pacemakers
* Participant whose circumstance is deemed by investigator to be unadvisable, unsafe, or unlikely to be capable of adhering to LCMR and/or isCGM/CBG monitoring during the study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who achieve remission at the end of phase 2 | from enrollment to end of phase 2 (18-30 weeks)
  The primary objective is to compare the percentage of participants who achieve remission of T2D (remission to prediabetes with HbA1c 6.0% to 6.4% or remission to normoglycemia with HbA1c < 6.0%) using no antihyperglycemic agents for ≥ 3 consecutive months at 18-30 weeks follow-up between isCGM vs. CBG monitoring, when combined with LCMR and DSME

SECONDARY OUTCOMES:
Proportion of participants achieving remission at the end of phase 1 | from enrollment to end of phase 1 (12-24 weeks)
  Evaluating the proportion of participants achieving remission of T2D (remission to prediabetes with HbA1c 6.0% to 6.4% or remission to normoglycemia with HbA1c < 6.0%) using no antihyperglycemic agents for ≥ 3 consecutive months at 12-24 weeks follow-up between intervention and control (isCGM vs. CBG monitoring, when combined with LCMR and DSME)
Proportion of participants achieving remission to prediabetes at the end of phase 1 | from enrollment to end of phase 1 (12-24 weeks)
  Evaluating the proportion of participants between intervention and control groups achieving remission to prediabetes (HbA1c 6.0% to 6.4%) using no antihyperglycemic agents for ≥ 3 consecutive months at weeks 12-24 weeks follow-up
Proportion of participants achieving remission to normoglycemia at the end of phase 1 | from enrollment to end of phase 1 (12-24 weeks)
  Evaluating the proportion of participants between the intervention and control group achieving remission to normoglycemia (HbA1c < 6.0%) using no antihyperglycemic agents for ≥ 3 consecutive months at weeks 12-24 weeks follow-up
Follow-up and change in HbA1c for the participants who did not initiate/reinitiate antihyperglycemic agents at the end of Phase 1 | from enrollment to end of Phase 1 (12-24 weeks)
  comparing between intervention and control (isCGM vs. CBG monitoring, when combined with LCMR and DSME) the follow-up HbA1c (%) and the change in HbA1c (%) at the end of Phase 1 (12-24 weeks) for participants who did not initiate/reinitiate antihyperglycemic agents
Adherence to low calorie meal replacement at the end of phase 1 | from enrollment to end of Phase 1 (12-24 weeks)
  Comparing the adherence to low calorie meal replacement (LCMR), defined as a score of 3, 4 or 5 out of 5 for LCMR adherence measured using the adherence questionnaire between the intervention and the control group at the end of phase 1 (12-24 weeks). A higher score on the scale indicates better adherence.
Percentage relapse at the end of Phase 1 | from enrollment to end of Phase 1 (12-24 weeks)
  comparing the number of participants between intervention and control group that relapse during Phase 1, reported as a percentage. Relapse is defined as weight gain > 2 kg from baseline body weight, HbA1c > 9%, fasting glucose > 11 mmol/L (on consecutive days, after first 4 weeks of LCMR), completely abandoning LCMR, and/or if participant needs to restart medications to lower their blood sugar (based on the doctor's recommendations).
Time spent in Phase 1 | from enrollment to end of phase 1 (12-24 weeks)
  Comparing the time spent in Phase 1 (12-24 weeks) between intervention and control group. Time spent will be measured in weeks
Proportion of participants achieving remission to prediabetes at the end of phase 2 | from enrollment to end of phase 2 (18-30 weeks)
  Evaluating the proportion of participants between intervention and control groups achieving remission to prediabetes (HbA1c 6.0% to 6.4%) using no antihyperglycemic agents for ≥ 3 consecutive months at 18-30 weeks follow-up
Proportion of participants achieving remission to normoglycemia at the end of phase 2 | from enrollment to end of phase 2 (18-30 weeks)
  Evaluating the proportion of participants between the intervention and control group achieving remission to normoglycemia (HbA1c < 6.0%) using no antihyperglycemic agents for ≥ 3 consecutive months at weeks 18-30 weeks follow-up
Follow-up and change of scores for Diabetes Treatment Satisfaction Questionnaire status version (DTSQs) scale at the end of phase 2 | from enrollment to end of phase 2 (18-30 weeks)
  Evaluating the follow-up and change in scores for the Diabetes Treatment Satisfaction Questionnaire status version (DTSQs) scale between the intervention and control group at the end of phase 2 ( 18-30 weeks). The DTSQs scale has 8 questions measured on a Likert scale from 6 (very satisfied) to 0 (very dissatisfied) about the participants satisfaction with their diabetes treatment in the last few weeks.
Follow-up and change in scores for the Diabetes Treatment Satisfaction Questionnaire change version (DTSQc) scale at the end of phase 2 | from enrollment to end of phase 2 (18-30 weeks)
  Evaluating the follow-up and change in scores for the Diabetes Treatment Satisfaction Questionnaire change version (DTSQc) scale between the intervention and control group at the end of phase 2 (18-30 weeks). The DTSQc scale has 8 questions measured on a Likert scale from 3 (much more satisfied now) to -3 (much less satisfied now) about the participants satisfaction of their diabetes treatment in the past 4-7 months.
Follow-up and change of scores in the Diabetes Distress scale (DDS) at the end of phase 2 | from enrollment to end of phase 2 (18-30 weeks)
  Evaluating the follow-up and change in scores in the Diabetes Distress scale (DDS) at the end of phase 2 (18-30 weeks) between intervention and control group. The DSS includes 17 questions measured on a Likert scale from 1 (not a problem) to 6 (a very serious problem) about the degree that diabetes has caused the participant distress in the past month. A higher score is reflective of more distress.
Proportion of participants achieving remission of T2D at the end of phase 3 | from enrollment to end of phase 3 (30-44 weeks)
  Evaluating the proportion of participants who achieve remission of T2D (remission to prediabetes with HbA1c 6.0% to 6.4% or remission to normoglycemia with HbA1c < 6.0% using no antihyperglycemic agents for ≥ 3 consecutive months) at 30-44 weeks follow-up between intervention and control ( isCGM vs. CBG monitoring, when combined with LCMR and DSME)
Proportion of participants achieving remission to prediabetes at the end of phase 3 | from enrollment to end of phase 3 (30-44 weeks)
  Evaluating the proportion of participants achieving remission to prediabetes (HbA1c 6.0% to 6.4% using no antihyperglycemic agents for ≥ 3 consecutive months) at 30-44 weeks between intervention and control group (isCGM vs. CBG monitoring, when combined with LCMR and DSME)
Proportion of participants achieving remission to normoglycemia at the end of phase 3 | from enrollment to end of phase 3 (30-44 weeks)
  Evaluating the proportion of participants achieving remission to normoglycemia (HbA1c < 6.0% using no antihyperglycemic agents for ≥ 3 consecutive months) at 30-44 weeks follow-up between intervention and control group ( isCGM vs. CBG monitoring, when combined with LCMR and DSME)
Evaluating the change in HbA1c at the end of phase 3 | from enrollment to end of phase 3 (30-42 weeks)
  Evaluating the change in HbA1c (%) at 30-44 weeks follow-up between intervention and control group
Low Calorie Meal Replacement persistence at the end of Phase 3 | End of Phase 3 (30-42 weeks)
  Comparing the persistence to Low Calorie Meal Replacement (LCMR) in percentage between the intervention and the control group at the end of phase 3 (30-44 weeks).
Proportion of participants initiating/reinitiating antihyperglycemic agents at the end of phase 3 | from enrollment to end of phase 3 ( 30-44 weeks)
  Evaluating the proportion of participants initiating/reinitiating antihyperglycemic agents at the end of phase 3 (30-44 weeks) between the intervention and control group.
Follow-up and change in body weight at the end of phase 3 | from enrollment to end of phase 3 (30-44 weeks)
  Evaluating the follow-up and change in body weight (kg) at the end of phase 3 (30-44 weeks) between the intervention and control group
Follow-up and change in BMI at the end of phase 3 | from enrollment to end of Phase 3 (30-44 weeks)
  Evaluating the follow-up and change in BMI (kg/m^2) at the end of phase 3 ( 30-44 weeks) between the intervention and control group
Percent weight loss at the end of Phase 3 | from enrollment to end of Phase 3 (30-44 weeks)
  Evaluating the percent weight loss at the end of Phase 3 (30-44 weeks) between the intervention and control group
Follow-up and change in scores for the Diabetes Treatment Satisfaction Questionnaire status version at the end of Phase 3 | from enrollment to end of Phase 3 ( 30-44 weeks)
  Evaluating the follow-up and change in scores for the Diabetes Treatment Satisfaction Questionnaire status version (DTSQs) between the intervention and control group at the end of phase 3 (30-44 weeks). The DTSQs scale has 8 questions measured on a Likert scale from 6 (very satisfied) to 0 (very dissatisfied) about the participants satisfaction with their diabetes treatment in the last few weeks.
Follow-up and change in scores in the Diabetes Distress scale (DDS) at the end of phase 3 | from enrollment to end of Phase 3 (30-44 weeks)
  Evaluating the follow-up and change in scores in the Diabetes Distress scale (DDS) at the end of phase 3 (30-44 weeks) between intervention and control group. The DSS includes 17 questions measured on a Likert scale from 1 (not a problem) to 6 (a very serious problem) about the degree that diabetes has caused the participant distress in the past month. A higher score is reflective of more distress
Change in Percent Time in Range (TIR) at the end of Phase 3 | from enrollment to end of Phase 3 (30-44 weeks)
  Evaluating the change in percent TIR (3.9 to 10.0 mmol/L) at the end of phase 3 (30-44 weeks) from baseline between intervention and control group
Change in Percent Tight Time in Range (TITR) at the end of Phase 3 | enrollment to end of Phase 3 (30-44 weeks)
  Evaluating the change in percent TITR (3.9 to 7.8 mmol/L) at the end of phase 3 (30-44 weeks) from baseline between intervention and control group
Change in Percent Time Below Range (TBR) at the end of Phase 3 | from enrollment to end of phase 3 (30-44 weeks)
  Evaluating the change in percent TBR (≤ 3.8 mmol/L) at the end of phase 3 (30-44 weeks) from baseline between intervention and control group
Change in Percent Time Below Range Level 1 at the end of Phase 3 | from enrollment to end of Phase 3 (30-44 weeks)
  Evaluating the change in percent TBR level 1 hypoglycemia range (3.0 to 3.8 mmol/L) at the end of phase 3 (30-44 weeks) from baseline between intervention and control group
Change in Percent Time Below Range Level 2 at the end of Phase 3 | from enrollment to end of Phase 3 (30-44 weeks)
  Evaluating the change in percent TBR level 2 hypoglycemia range (< 3.0 mmol/L)at the end of phase 3 (30-44 weeks) from baseline between intervention and control group
Change in Percent Time Above Range (TAR) at the end of Phase 3 | from enrollment to end of Phase 3
  Evaluating the change in percent TAR (> 10.0 mmol/L) at the end of phase 3 (30-44 weeks) from baseline between intervention and control group
Change in mean glucose at the end of Phase 3 | from enrollment to end of Phase 3 (30-44 weeks)
  Evaluating the change in mean glucose (mmol/L) at the end of phase 3 (30-44 weeks) from baseline between the intervention and control group.
Change in Glycemic Variability at the end of Phase 3 | from enrollment to end of Phase 3 (30-44 weeks)
  Evaluating change in glycemic variability (standard deviation and % coefficient of variation) from baseline to the end of Phase 3 (30-44 weeks) between the intervention and control group.
Change in Glucose Management Indicator at the end of Phase 3 | from enrollment to end of Phase 3 (30-44 weeks)
  Evaluating the change in Glucose management indicator, measured in percentage (%) between the intervention and control group from baseline to the end of Phase 3 (30-44 weeks)

OTHER OUTCOMES:
Evaluating isCGM metrics at the end of phase 3 between isCGM+ LCMR+ DSME and CBG+ LMCR+ DSME | End of Phase 3 (30-44 weeks)
  Evaluating isCGM metrics (collected from a blinded isCGM) between isCGM vs. CBG monitoring, when combined with LCMR and DSME at 30-42 weeks follow-up. We will describe the mean (SD) and/or median (IQR) for TIR and TITR among the pooled sample of participants from both randomized arms (isCGM and CBG) achieving remission to prediabetes or remission to normoglycemia.

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (6):
  - LMC Brampton, Brampton, Ontario
  - LMC Etobicoke, Etobicoke, Ontario
  - LMC Oakville, Oakville, Ontario
  - LMC Ottawa, Ottawa, Ontario
  - LMC Bayview, Toronto, Ontario
  - LMC Vaughan, Vaughan, Ontario

IPD SHARING:
Plan to Share IPD: No